CLINICAL TRIAL: NCT06098742
Title: An Open-label, Randomized, Crossover Study to Investigate the Comparative Pharmacodynamics and Pharmacodynamics Equivalence of Antareit 800 mg/10 ml Oral Suspension and Riopan 800 mg Chewable Tablets in Healthy Volunteers.
Brief Title: Comparative Pharmacodynamics and Pharmacodynamics Equivalence of Antareit 800 mg/10 ml Oral Suspension and Riopan 800 mg Chewable Tablets in Healthy Volunteers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ANT-05-01-2022
Record Dates: First submitted 2023-10-19; First posted 2023-10-24 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Heartburn; Acid-dependent Diseases of the Gastrointestinal Tract; Symptomatic Treatment of Gastric and Duodenal Ulcers
MeSH Terms: conditions — Heartburn; Duodenal Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TR-sequence (T-test drug, R-reference drug) (Experimental): Group 1 (25 volunteers, TR sequence) will take 2 sachets of Antareit 800 mg/10 ml oral suspension 2 h prior to food intake in Period 1 and 2 tablets of Riopan 800 mg chewable tablets 2 h prior to food intake in Period 2
  Interventions: Drug: Antareit
- RT-sequence (Experimental): Group 2 (25 volunteers, RT sequence) will take 2 tablets of Riopan 800 mg chewable tablets 2 h prior to food intake in Period 1 and 2 sachets of Antareit 800 mg/10 ml oral suspension 2 h prior to food intake in Period 2
  Interventions: Drug: Antareit

INTERVENTIONS:
Drug: Antareit — A single dose of T or R drug in each of 2 periods of the study 2 h prior to food intake

SUMMARY:
Comparative study of the pharmacodynamic parameters and pharmacodynamic equivalence (bioequivalence) of drug Antareit 800 mg/10 ml oral suspension and drug Riopan 800 mg chewable tablets in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary and handwritten informed consent form signed by a healthy volunteer to participate in the study prior to any of the study procedures;
2. Healthy male and female caucasian volunteers aged 18 to 45 years (inclusive);
3. Verified diagnosis "healthy" (without abnormal findings in the protocol-defined clinical, laboratory, and instrumental test data);
4. pH according to hourly pH-metry in the screening period, carried out at least 3 hours after the last meal, is completely in the range from 1 to 3 inclusive throughout the entire astronomical hour of measurement;
5. Blood pressure (BP) levels: 100 to 139 mm Hg, inclusive (systolic, SBP), 60 to 89 mm Hg, inclusive (diastolic, DBP);
6. Heart rate (HR) of 60 to 90 bpm, inclusive;
7. Body mass index (BMI) of 18.5 kg/m2 ≤ BMI ≤ 30 kg/m2, where the body weight range is ≥ 55 kg for men and ≥ 45 kg for women;
8. Non-smoking healthy volunteers (who have never smoked or gave up smoking more than 6 months prior to the Screening);
9. Consent to use adequate methods of contraception throughout the study and for 30 days after completion; for women of preserved reproductive potential, a negative urine pregnancy test result;
10. The volunteers must have adequate behavior and coherent speech.

Exclusion Criteria:

1. A history of allergy;
2. History of drug intolerance to the active and/or excipients included in the study drugs;
3. History of drug intolerance of or hypersensitivity/allergic reactions to lidocaine, xylocaine or other topical anesthetics which will be used at the trial site for anesthesia during esophagogastroduodenoscopy (EGD) and insertion of the probe for the pH measurements;
4. Chronic diseases of the circulatory, lymphatic, respiratory, nervous, endocrine, gastrointestinal, musculoskeletal, integumentary, immune, urogenital, and hematopoietic systems;
5. Esophageal, gastric, and/or duodenal diseases based on EGC performed at screening and based on the medical history; a history of esophageal, gastric, and/or duodenal surgery;
6. Diseases/conditions which, in the opinion of the investigator, may affect the pH measurement results;
7. Acute infectious diseases less than 4 weeks prior to screening;
8. Use of antacids (including sodium bicarbonate solution)/H2 antagonists 24 h prior to the Screening Visit;
9. Use of proton pump inhibitors 72 h prior to the Screening Visit;
10. Use of (including use of a single dose) steroids and/or other ulcerogenic drug (e.g., nonsteriodal anti-inflammatory drugs [NSAID]) less than 4 weeks prior to the Screening Visit;
11. Regular use of any medicinal products, including prescription only and OTC (Over-the-counter) drugs and dietary supplements within 2 weeks prior to the Screening Visit;
12. Blood or plasma donation less than 3 months prior to the Screening Visit;
13. Use of hormonal contraceptives (in women) less than 2 months prior to the Screening Visit;
14. Pregnancy or breastfeeding; a positive pregnancy test for women of childbearing potential;
15. Participation in another clinical trial less than 3 months prior to screening or simultaneously with this study;
16. Use of more than 10 units of alcohol (1 unit of alcohol is equivalent to 330 ml of beer, 150 ml of wine or 40 ml of spirits) a week within a month prior to the enrollment in the study or history data of alcohol/drug dependence or drug abuse.
17. Positive antibody blood test for HIV-1 and HIV-2, Treponema pallidum antigen, hepatitis B surface antigen (HBsAg), or hepatitis C virus antigen;
18. Positive urine test for narcotic substances or strong drugs;
19. Positive test for alcohol vapor in exhaled breath or a positive alcohol saliva test;
20. Deviated septum/nasal obstruction preventing the placement of the pH probe;
21. Medical history of chronic constipation;
22. Medical history of severe maxillofacial injuries;
23. Expected admission to hospital during this study for any reason, except for hospitalization provided for by this protocol;
24. Impossibility or failure to comply with the protocol, undergo protocol-defined procedures, or adhere to the diet or activity regime;
25. Positive SARS-CoV-2 (severe acute respiratory syndrome related coronavirus) (COVID-19) rapid test;
26. Other circumstances which in the opinion of the investigator prevent a volunteer from being included in the study or may result in premature drop-out from the study.

Withdrawal criteria:

1. The volunteer's refusal to further participate in the study;
2. Failure of the volunteer to comply with the rules of participation in the study (skipping study procedures, independent use of drugs prohibited in the study, violation of dietary and lifestyle restrictions, etc.);
3. Taking prohibited therapy;
4. Occurrence of causes/occurrence during the study of situations that threaten the safety of the volunteer, including severe AEs;
5. Volunteers selected to participate in the study in violation of the inclusion/non-inclusion criteria;
6. Violation of the rules for conducting pH measurements or the occurrence of conditions that required early termination of pH measurements (vomiting, nosebleeds, etc.);
7. Missing a dose of the study drug/comparator drug during any period of the study for any reason;
8. Positive urine test for narcotics and powerful drugs;
9. Positive breath alcohol vapor test or alcohol in saliva;
10. Positive pregnancy test in women;
11. Positive test for COVID-19;
12. The occurrence in the course of the study of other reasons that prevent the study according to the protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-10-20 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Pharmacodynamics - AUCpH - Area under the curve potential of hydrogen | From 0 to 1 hour (Day 1 and Day 8)
  Area under the pharmacodynamic pH-time curve
Pharmacodynamics - time percentage during which the intragastric pH value will exceed 4.0 | From 0 to 1 hour (Day 1 and Day 8)
  PH - potential of hydrogen
Pharmacodynamics- рНmaximum | From 0 to 1 hour (Day 1 and Day 8)
  maximum potential of hydrogen
Pharmacodynamics- рНmin | From 0 to 1 hour (Day 1 and Day 8)
  minimum potential of hydrogen
Pharmacodynamics - average pH value | From 0 to 1 hour (Day 1 and Day 8)
  root mean square
Pharmacodynamics - time percentage during which the intragastric pH value will exceed 3.0 | From 0 to 1 hour (Day 1 and Day 8)
  During which the intragastric pH value will exceed 3.0
Pharmacodynamics - median time when the pH was above 3.0 | From 0 to 1 hour (Day 1 and Day 8)
Pharmacodynamics - median time when the pH was above 4.0 | From 0 to 1 hour (Day 1 and Day 8)

SECONDARY OUTCOMES:
Safety and Tolerability: adverse event (AE) number and frequency | From the screening (and signing informed consent form) to Day 15 of the study or to an early termination visit within the time frame of the study (from Day 0 to Day 15)
  Number and frequency of adverse events (AEs) or serious AEs (SAEs)
Safety and Tolerability: serious adverse event (SAE) number and frequency | From the screening (and signing informed consent form) to Day 15 of the study or to an early termination visit within the time frame of the study (from Day 0 to Day 15)
  Number and frequency of serious AEs (SAEs)
Safety and Tolerability: volunteer complaints | From the screening (and signing informed consent form) to Day 15 of the study or to an early termination visit within the time frame of the study (from Day 0 to Day 15)
Safety and Tolerability: physical examination results | Screening, from Day 0 to Day 2, from Day 7 to Day 9, and/or on early termination visit within the time frame of the study (from Day 0 to Day 15)
  Physical examination will be conducted to identify normal and abnormal physical characteristics of volunteers in accordance with the planned examination and will include an assessment of the Condition of the cardiovascular, respiratory, digestive, endocrine, musculoskeletal, nervous, sensory systems, skin/visible mucous membranes
Safety and Tolerability: vital signs | Screening, from Day 0 to Day 2, from Day 7 to Day 9, and/or on early termination visit within the time frame of the study (from Day 0 to Day 15)
  systolic blood pressure (SBP),diastolic blood pressure (DBP), heart rate (HR), body temperature
Safety and Tolerability: 12-lead electrocardiogram (ECG) | Screening, Day 9
  12-lead ECG (I, II, III, aVR -enhanced unipolar abduction from the right arm , aVL - enhanced unipolar abduction from the left arm , aVF - enhanced unipolar abduction from the left legб V1-V6) taken while lying down: heart rate (beats per minute), PQ interval (is the period, measured in milliseconds, that extends from the beginning of the P wave (the onset of atrial depolarization) until the beginning of the QRS complex), QRS complex (The QRS complex is the combination of three of the graphical deflections seen on a typical electrocardiogram), corrected QT interval (distance from the beginning of the QRS complex to the end of the T wave)
Safety and Tolerability: clinical blood test | Screening, Day 2, Day 9
  hemoglobin, hematocrit, Red blood cell count, Platelet count, Leukocyte count, erythrocyte sedimentation rate, Leukocyte formula (myelocytes, band neutrophils, segmented neutrophils, eosinophils, basophils, monocytes, lymphocytes)
Safety and Tolerability: blood chemistry | Screening, Day 2, Day 9
  Glucose concentration, Total cholesterol concentration, Total protein concentration, Total bilirubin concentration, Creatinine concentration, Alkaline phosphatase activity, alanine transaminase and aspartate transaminase activity
Safety and Tolerability: urinalysis | Screening, Day 2, Day 9
  Relative density, Color, Transparency, pH, Protein concentration, Glucose concentration, Red blood cell content, White blood cell content, Epithelial cell content, Presence of casts, Presence of mucus, Presence of bacteria.
Safety and Tolerability: urinalysis (microscopy) | Screening, Day 2, Day 9
  Microscopy of urine sediment is performed if it is present.

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Llc "Certa Clinic", Moscow
  - Limited Liability Company "Research Center Eco-Safety", Saint Petersburg

IPD SHARING:
Plan to Share IPD: Undecided